CLINICAL TRIAL: NCT04532489
Title: Positron Emission Tomography (PET) Imaging of Cholesterol Trafficking: Clinical Evaluation of [18F]FNP-59 in Normal Human Subjects (Group 1)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benjamin Viglianti (Other)
Responsible Party: Sponsor-Investigator, Benjamin Viglianti, Assistant Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00179097a
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Radiotracer; Hypertension; Cholesterol
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Other): These subjects, 6 planned (3 male, 3 female), will be to obtain normal tissue distribution of [18F]NP-59 and confirm calculated radiation dosimetry and optimal uptake time.
  Interventions: Drug: FNP-59

INTERVENTIONS:
Drug: FNP-59 — FNP-59, a radiotracer, is administered for PET/CT scans.

SUMMARY:
This exploratory, first-in-man, phase 0 study will evaluate the feasibility of using a sub-therapeutic dose of a fluorine-18 analogue of NP-59 ([18F]FNP-59) to image the adrenal gland in healthy normal subjects. The researchers believe that [18F]FNP-59 would greatly improve the imaging characteristics, by providing a PET imaging cholesterol analogue with significantly improved radiation dosimetry.

DETAILED DESCRIPTION:
Following the results of radiation dosimetry from this study then next steps will be taken for groups 2 & 3 using hormone manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Participants without any known adrenal pathology as normal controls for radiation dosimetry purposes

Exclusion Criteria:

* Pregnancy
* Unable to do imaging
* Body weight greater than 400 lbs (181 Kg)
* Prisoners are not eligible
* Subjects unable to provide own consent are not eligible
* Current use of steroids, Oral contraceptives (OCP), spironolactone, estrogen, androgen, progesterone, Angiotensin-converting enzyme (ACE inhibitors)/ Angiotensin II receptor blockers (ARBs), or supplements that are hormone analogues.
* Known adrenal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Uptake for [18F]FNP-59 in the adrenal glands using the standardized uptake value (SUV) based on gland segmentation | Day 0
  SUV will be reported. Both maximal and average SUVs will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ben Viglianti, M.D, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No